CLINICAL TRIAL: NCT00876122
Title: An Open-Label, Phase I, Dose-Escalation Study of PI3-Kinase Inhibitor (GDC-0941) in Patients With Locally Advanced or Metastatic Solid Tumors or Non-Hodgkin's Lymphoma for Which Standard Therapy Either Does Not Exist or Has Proven Ineffective or Intolerable
Brief Title: A Study of GDC-0941 in Patients With Locally Advanced or Metastatic Solid Tumors or Non-Hodgkin's Lymphoma for Which Standard Therapy Either Does Not Exist or Has Proven Ineffective or Intolerable
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDC4254g; GO01299 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-03-13; First posted 2009-04-06 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Non-Hodgkin's Lymphoma, Solid Cancers
Keywords: NHL; Metastatic Solid Tumors; PI3K Inhibitors; PI3K
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — 2-(1H-indazol-4-yl)-6-(4-methanesulfonylpiperazin-1-ylmethyl)-4-morpholin-4-ylthieno(3,2-d)pyrimidine

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: GDC-0941

INTERVENTIONS:
Drug: GDC-0941 — Escalating oral dose

SUMMARY:
This is an open-label, Phase I, dose-escalation study using a 3 + 3 design to assess the safety, tolerability, and pharmacokinetics of orally administered GDC-0941 administered QD. This study will include patients with locally advanced or metastatic solid tumors, NHL, or multiple myeloma (MM) (expansion stage only) for which standard therapy either does not exist or has proven ineffective or intolerable.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented, incurable, locally advanced or metastatic solid malignancy or NHL without leukemic phase that has progressed or has failed to respond to at least one prior regimen
* Multiple myeloma (MM) patients (only in Stage 2): documented pathologic diagnosis of MM that has relapsed or that has failed to respond after treatment with at least one prior systemic therapy (other than corticosteroid monotherapy)
* Evaluable or measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) or per International Working Group (IWG) response criteria for Non-Hodgkin's lymphoma (NHL) patients
* Life expectancy of >= 12 weeks
* Documented willingness to use an effective means of contraception for both men and women while participating in the study
* For patients participating in Stage 1 after an adequate exposure has been predicted or observed on the basis of PK analysis and for approximately 12 patients participating in Stage 2 (excluding patients with MM): A biopsy-accessible lesion from which tissue can be obtained safely with CT guidance or direct visualization and agreement from the patient to undergo sequential (pre-treatment and post-treatment) biopsies.
* For patients participating in Stage 2 DCE-MRI and MRS imaging: Patients will have at least one metastatic liver lesion measuring >= 5 cm in one dimension or one tumor lesion elsewhere measuring >= 2 cm in one dimension (lung and mediastinum lesions do not qualify) on the basis of CT scans

Exclusion Criteria:

* Leptomeningeal disease as the only manifestation of the current malignancy
* History of Type 1 or 2 diabetes mellitus requiring regular medication
* Any condition requiring anti-coagulants, such as warfarin, heparin, or thrombolytics
* Inability or unwillingness to swallow pills
* Malabsorption syndrome or other condition that would interfere with enteral absorption
* Known untreated CNS malignancies or treated brain metastases that are not radiographically stable for >= 3 months
* Congenital long QT syndrome or QTc > 500 msec, as determined by at least two of the three baseline ECG measurements
* Active congestive heart failure or ventricular arrhythmia requiring medication
* Uncontrolled ascites requiring weekly large volume paracentesis for 3 consecutive weeks prior to enrollment
* Active infection requiring intravenous (IV) antibiotics
* Patients requiring any daily supplemental oxygen
* DLco, 50% predicted value corrected for AV and Hgb prior to initiation of study treatment
* Uncontrolled hypomagnesemia or hypokalemia, defined as values below the lower limit of normal (LLN) or hypercalcemia above the ULN for the institution despite adequate electrolyte supplementation or management
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Known human immunodeficiency virus (HIV) infection
* Any other diseases, active or uncontrolled pulmonary dysfunction, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or renders the patients at high risk from treatment complications
* Significant traumatic injury within 3 weeks before Day 1
* Major surgical procedure within 4 weeks prior to initiation of study treatment
* Prior allogeneic hematopoietic stem cell transplantation (HSCT) at any time or autologous HSCT within 12 weeks of study entry
* Treatment with chemotherapy, hormonal therapy (except GnRH agonists or antagonists for prostate cancer), immunotherapy, biologic therapy, or radiation therapy (except palliative radiation to bony metastases) as cancer therapy within 4 weeks prior to initiation of study treatment (exceptions are kinase inhibitors that are approved by the local regulatory authorities, which may be used within 2 weeks prior to initiation of study treatment, provided that any drug-related toxicity has completely resolved and after approval by the Medical Monitor has been granted)
* Palliative radiation to bony metastases within 2 weeks prior to initiation of study treatment
* Need for chronic corticosteroid therapy
* Treatment with an investigational agent within 4 weeks prior to initiation of study treatment
* Unresolved toxicity from prior therapy, except for alopecia and Grade 1 peripheral neuropathy
* Pregnancy or lactation
* Inability to comply with study and follow-up procedures
* For patients eligible to participate in Stage 2 DCE-MRI and MRS assessments, any contraindication to MRI examination, including the following:

Imbedded metallic material/devices (metal implants or large tattoos in the field of view)

Severe claustrophobia

Physical characteristics (weight or size) that exceed the capabilities of the MRI scanner

Known allergy or hypersensitivity reactions to gadolinium, verse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events by NCI CTCAE grade and associated dose of GDC-0941 | Through study completion or early study discontinuation
Occurrence of dose-limiting toxicities (DLTs) by NCI CTCAE grade and associated dose of GDC-0941 | Through study completion or early study discontinuation
Occurrence of Grade 3 or 4 abnormalities in safety-related laboratory parameters and associated dose of GDC-0941 | Through study completion or early study discontinuation
PK parameters after single and multiple doses of GDC-0941 | Through study completion or early study discontinuation

SECONDARY OUTCOMES:
Positron emission tomography (PET) response for patients with detectable FDG tumor uptake at baseline | Through study completion or early study discontinuation
Best overall response, duration of objective response, and progression-free survival (PFS) for patients with measurable disease according to RECIST | Through study completion or early study discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Gallia Levy, M.D., Study Director — Genentech, Inc.
Locations (1):
- Sutton, United Kingdom